CLINICAL TRIAL: NCT07336368
Title: Topical Cryotherapy to Reduce Pain During Steroid Injections for Keloid and Hypertrophic Scars: A Pilot Study
Brief Title: Topical Cryotherapy and Keloid/Hypertrophic Scars
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sonal Choudhary (Other)
Responsible Party: Sponsor-Investigator, Sonal Choudhary, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY25080173
Record Dates: First submitted 2026-01-10; First posted 2026-01-13 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Keloid Scars; Hypertrophic Scars
Keywords: Keloid scars; Hypertrophic scars; Cryotherapy; Intralesional corticosteroids; Pain reduction; Injection resistance; Injection pain
MeSH Terms: conditions — Keloid; Cicatrix, Hypertrophic | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cryotherapy + Steroids vs Steroids alone (Experimental): A provider will divide the identified keloid into two halves. The division will be marked down the center using a sterile skin marker under standard aseptic conditions. The provider will then administer the intervention; one half of the keloid will receive cryoanesthesia with liquid nitrogen spray (~10 seconds). Within the next 60 seconds, standard intralesional triamcinolone (10-40 mg/mL) will be injected in that half using an identical needle gauge, depth, and volume planned for clinical care. The other half will receive standard intralesional triamcinolone only with an identical injection technique and dose.
  Interventions: Device: Cryotherapy with liquid nitrogen; Drug: Intralesional Triamcinolone 10 mg/ml

INTERVENTIONS:
Device: Cryotherapy with liquid nitrogen — liquid nitrogen spray (~10 seconds)
Drug: Intralesional Triamcinolone 10 mg/ml — Intralesional triamcinolone

SUMMARY:
The goal of this clinical trial is to determine whether the application of brief topical cryotherapy immediately before intralesional corticosteroid injections can reduce pain and injection resistance during routine treatment of keloid and hypertrophic scars in adult patients.

The main questions it aims to answer are:

Does topical cryotherapy applied before intralesional triamcinolone injection impact pain perceptions for participants with keloids or hypertrophic scars?

Does topical cryotherapy affect provider-assessed injection resistance compared with standard injection alone?

Researchers will split the keloid/hypertrophic scar into two halves. One half will be treated with cryotherapy followed by steroid injection, while the other half will be treated with steroid injection alone to evaluate differences in pain perception and injection resistance.

Participants will rate pain after each injection using a 10-point numeric pain scale. Clinicians will rate the resistance after each injection using a 10-point numeric scale.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with keloids or hypertrophic scars already scheduled to receive intralesional triamcinolone (TAC) as part of routine care.
* At least one keloid or hypertrophic scar with two comparable regions (≥2 cm each) suitable for split-treatment.
* Able to provide informed consent and complete pain assessments in English.

Exclusion Criteria:

* Keloid or hypertrophic scar located on the face (except earlobes), excluded for cosmetic reasons.
* Prior treatment to the study-selected keloid/hypertrophic scar based on self-report.
* Inability to complete study assessments due to cognitive or language barriers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Patient pain perceptions | Immediately following intralesional corticosteroid injection (same visit)
  Pain perception during intralesional corticosteroid injection will be assessed using a patient-reported numeric rating scale (0 = No pain, 10 = Very severe pain).
Provider-reported resistance of injection | Immediately following intralesional corticosteroid injection (same visit)
  Dermatology providers will rate resistance of the intralesional corticosteroid injection using a 10-point numeric scale (0 = No resistance to 10 = Very strong resistance).

CONTACTS AND LOCATIONS:
Overall Officials: Sonal Choudhary, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data will not be shared to protect participants' privacy; only aggregate results will be reported.